CLINICAL TRIAL: NCT03972072
Title: MARTHA-trial: MRI - Guided Adaptive RadioTHerapy for Reducing XerostomiA in Head and Neck Cancer Including Longitudinal Evaluation of the Patient's Immune Profile Under Radiotherapy
Brief Title: MRI - Guided Adaptive RadioTHerapy for Reducing XerostomiA in Head and Neck Cancer (MARTHA-trial)
Acronym: MARTHA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Panagiotis Balermpas (Other)
Responsible Party: Sponsor-Investigator, Panagiotis Balermpas, Sponsor-Investigator, Senior Consultant, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN01_2019
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer; Xerostomia Due to Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Intervention Arm (Experimental): daily imaging for MR-IGRT once weekly offline plan adaptation subjective/objective LENT-SOMA xerostomia-evaluation including flow measurements at baseline, 6 month-, 12 month- and 24 month-follow up EORTC-QoL questionnaires at baseline, 6 month-, 12 month- and 24 month-follow up
  Interventions: Other: Pre-defined MR-linac based IGRT and plan adaptation protocol; Diagnostic Test: salivary flow measurements

INTERVENTIONS:
Other: Pre-defined MR-linac based IGRT and plan adaptation protocol — daily MR-imaging/MR guided radiotherapy once weekly offline plan adaptation to a total of 6
Diagnostic Test: salivary flow measurements — baseline, 6 month-, 12 month- and 24 month-follow up salivary flow measurements and LENT-SOMA subjective/objective evaluation of xerostomia

SUMMARY:
Radiotherapy is the main treatment for locally advanced squamous cell carcinoma of the head and neck (SCCHN). Many advances regarding tumor control and patient survival have been made over the past decades. However, treatment-induced toxicity remains a crucial problem, leading to reduced quality of life and permanent impairment for many survivors. Xerostomia is up to this day the leading cause of late toxicity for these patients. Toxicity has been reduced by implementation of modern image guided radiotherapy (IGRT) and intensity-modulated radiotherapy (IMRT), but the low soft-tissue contrast of routine x-ray image guidance does not allow exact planning adaptation and daily imaging is associated with high radiation exposure. Furthermore, despite the routinely use of IMRT, rates of clinically relevant xerostomia (i.e. grade 2 or worse) are still common and reported in approximately 38%. Recently developed hybrid machines (MRidian®-CE approval since 2016), consisting of a linear accelerator and an integrated low-field MRI, could allow a) better visualization of tumor and organs at risk, such as parotid glands during patient positioning and daily treatment, b) daily imaging without additional radiation exposure, c) narrowest established safety margins for the treatment volumes, and finally d) repetitive adaptation of target volumes according to changes in patient weight and tumor anatomy during the radiotherapy course. These procedures would facilitate a high-precision treatment and help reduce dose exposure of critical structures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the oral cavity oro- or hypopharynx or larynx, Stages II-IVB, requiring definitive or postoperative bilateral neck irradiation
* Age ≥ 18 years, no upper age limit
* ECOG-Performance score < 2
* The trial is open to both genders
* History/physical examination within 30 days prior to registration by head and neck surgeon and Radiation Oncologist
* FDG-PET-CT-scan within 30 days prior to registration

Exclusion Criteria:

* Not adequately controlled hepatitis or HIV disease (HIV-viral load detectable)
* Second non-controlled malignancy other than basalioma or cervical/genital/anal in situ neoplasia during the last 2 years before enrollment
* Bilirubin > 2,0 mg/dl, SGOT, SGPT, AP, Gamma-GT >3x norm, GFR < 30 ml/min
* leucocytes <3,5 x 10^9/l or platelets < 100 x 10^9/l or neutrophiles < 1,5 x 10^9/l
* Other severe comorbidities or psychic disorders (e.g. myocardial infraction within 6 months prior to registration, permanent cardiac arrhythmia, COPD Gold IV, hepatitis B/C, schizophrenia, ongoing alcohol abuse etc.)
* Lactating and pregnant women
* Previous radiotherapy of the neck
* Contraindications for MRI (e.g. pacemaker/ICD, tattoos, cochlear or other not MR-compatible implants)
* Pre-existing salivary gland disease (e.g. Sjorgen's-syndrome) or xerostomia-inducing medication (e.g. anticholinergic medication like tricyclic antidepressant)
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-05-21 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with xerostomia of grade 2 or worse | 12 month-follow up
  will be evaluated by the LENT-SOMA (Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA)) side-effect scale: SOM (1)-(4) (higher score represents higher grade xerostomia), A: objective flow measurement (1) 76-95%, (2) 51-75%, (3) 26-50%, (4) 0-25%

SECONDARY OUTCOMES:
Percentage of patients with xerostomia of grade 2 or worse | 6- and 24-months follow up
  will be evaluated by the LENT-SOMA (Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA)) side-effect scale: SOM (1)-(4) (higher score represents higher grade xerostomia), A: objective flow measurement (1) 76-95%, (2) 51-75%, (3) 26-50%, (4) 0-25%
Locoregional control rate as defined from treatment start to histologically confirmed tumor progression, persistence or last follow up | 2-years
  as defined from treatment start to histologically confirmed tumor progression, persistence or last follow up
Overall survival | 2-years
  as defined from treatment start to death from any cause or last follow up
Description of Quality of life - scoring 6 months after treatment, assessed according to the general EORTC-quality of life "core" questionnaire QLQ C30 (overall quality of life for cancer patients) | 6 months after treatment
  Questionnaire consists of 30 questions with a maximal score of 100. Absolute scores after linear transformation will be reported as descriptive statistics The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  See also: https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf
Description of Head-Neck cancer related symptoms 6 months after treatment, assessed according to the specific EORT-head and neck quality of life supplementary questionnaire HN35 | 6 months after treatment
  total scoring of an additional 35 questions with a similar approach to that of the core questionnaire will be reported as descriptive statistics
Description of Quality of life - scoring 12 months after treatment, assessed according to the general EORTC-quality of life "core" questionnaire QLQ C30 (overall quality of life for cancer patients) | 12 months after treatment
  Questionnaire consists of 30 questions with a maximal score of 100. Absolute scores after linear transformation will be reported as descriptive statistics The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  See also: https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf
Description of Head-Neck related symptoms 12 months after treatment, assessed according to the specific EORT-head and neck quality of life supplementary questionnaire HN35 | 12 months after treatment
  total scoring of an additional 35 questions with a similar approach to that of the core questionnaire will be reported as descriptive statistics
Description of Quality of life - scoring 24 months after treatment, assessed according to the general EORTC-quality of life "core" questionnaire QLQ C30 (overall quality of life for cancer patients) | 24 months after treatment
  Questionnaire consists of 30 questions with a maximal score of 100. Absolute scores after linear transformation will be reported as descriptive statistics The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  See also: https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf
Description of Head-Neck related symptoms 24 months after treatment, assessed according to the specific EORT-head and neck quality of life supplementary questionnaire HN35 | 24 months after treatment
  total scoring of an additional 35 questions with a similar approach to that of the core questionnaire will be reported as descriptive statistics
Toxicity rates | weekly during radiotherapy and at 3, 6, 9, 12, 15, 18, 21 and 24 months
  evaluated by the CTCAE v5-questionnaires

OTHER OUTCOMES:
variation of radiomics features (delta radiomics) of the parotid glands | Up to 9 weeks after enrollment: Images acquired at baseline (i.e. up to 10 days before first radiotherapy fraction, used for radiotherapy planning) and daily radiotherapy treatment (treatment days 1-35, 7 weeks)
  as assessed by serial T1/T2 images acquired with the hybrid 0.35 T MR-linac and correlated with xerostomia at 12 months
variation of tumor radiomics features (delta radiomics) for tumor control for the definitively irradiated (non-surgically treated) patients | Up to 9 weeks after enrollment: Images acquired at baseline (i.e. up to 10 days before first radiotherapy fraction, used for radiotherapy planning) and daily radiotherapy treatment (treatment days 1-35, 7 weeks)
  as assessed by serial T1/T2 images acquired with the hybrid 0.35 T MR-linac and correlated with tumor control at 24 months
longitudinal inflammation profiling | Up to 3 months after enrollment (value assessment at baseline, after one week of treatment, last week of treatment and first follow up)
  Prognostic value of inflammation surrogates (neutrophile count, CRP/ albumin ratio) in the peripheral blood
longitudinal immune profiling | Up to 3 months after enrollment (value assessment at baseline, after one week of treatment and first follow up)
  Prognostic value of different circulating (at different time-points) immune cells as defined by longitudinal FACS-analysis of immune phenotype in the peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Balermpas, M.D., Principal Investigator — University Hospital Zurich, Department of Radiation-Oncology
Locations (1):
- Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided